CLINICAL TRIAL: NCT02879721
Title: The Renin-angiotensin System (RAS) in Barrett's Esophagus as Future Biomarkers for Dysplasia and Cancer? A Randomized Controlled Trial
Brief Title: Expression and Function of the Renin-Angiotensin System in the Esophagus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 233-09
Record Dates: First submitted 2016-05-31; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Barrett's Esophagus
Keywords: Gastrointestinal
MeSH Terms: conditions — Barrett Esophagus | interventions — candesartan; candesartan cilexetil; Enalapril; Enalaprilat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- no drug (No Intervention): No drug and no intervention
- AT1R-antagonist (Active Comparator): Angiotensin II, type 1 receptor inhibitor, (candesartan) 8 mg once daily
  Interventions: Drug: Candesartan
- ACE-inhibitor (Active Comparator): Angiotensin converting enzyme inhibitor, (enalapril) 5 mg once daily
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Candesartan — Angiotensin II, type 1 receptor inhibitor, (candesartan) 8 mg once daily for
  Other Names: Atacand, Ratacand, Biopress; CAS 139481-59-7, ATC C09CA06
  Arms: AT1R-antagonist
Drug: Enalapril — Angiotensin-converting enzyme (ACE) inhibitor (enalapril) 5 mg once daily
  Other Names: Vasotec, Enaladex, Renitec; CAS 75847-73-3, ATC C09AA02
  Arms: ACE-inhibitor

SUMMARY:
Barrett's esophagus (BE) is the major esophageal pre-neoplastic lesion in which dysplastic transformations eventually can lead to cancer development. Today, the only way for early detection of pre-neoplastic lesions is an endoscopic surveillance programme with tissue sampling for histopathology, the latter being the only validated biomarker for esophageal adenocarcinoma (EAC)-risk available. New biomarkers are warranted for better patient selection before inclusion into BE surveillance programmes.

Epidemiologic studies have demonstrated suppressed numbers of cancer prevalence in cohorts being under different medical treatment. In a British epidemiological study 2007 Sjöberg et al noted a lower prevalence of EAC among patients treated with antihypertensive drugs interfering with the renin-angiotensin system (RAS) such as AT1R-blockers and ACE-inhibitors. The last decade this endocrine signalling system has been proven to be involved in pathological conditions such as inflammation, wound-healing and even cancer, in several organ systems.

Earlier reports from the investigators laboratory indicate the existence of a local RAS in the esophageal wall musculature and in the squamous mucosa. In the investigators latest explorative study, the investigators discovered the altered expression of "classical" RAS components in BE with and without dysplasia (unpublished results).

By a possible alteration in RAS-related protein-expression in BE with increasing grade of dysplasia towards EAC, the investigator may have a possible "pathway" leading to biomarkers for cancer-development. Furthermore, the already well-known anti-hypertensive drugs ACE-inhibitors and AT1R-blockers may interfere with the risk of malignancy in BE. The investigators therefore wish to test, in an exploratory prospective randomized placebo-controlled setting, whether RAS-related protein-expressions in BE are altered by the addition of RAS-suppressant pharmaceuticals. In the same manner the investigators wish to see if the expressions of well-known biomarkers for cancer and inflammation are altered.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is the major esophageal pre-neoplastic lesion in which dysplastic transformations eventually can lead to cancer development. Early detection of high-grade dysplasia (HGD) or intramucosal cancer is of fundamental value for the patient. The minimally invasive endoscopic resection- and ablation-techniques available are curative. In patients with invasive cancer far more invasive resection-techniques are required which are associated with severe post-operative morbidity, mortality and poor overall survival. Today, the only way for early detection of pre-neoplastic lesions is an endoscopic surveillance programme with tissue sampling for histopathology, the latter being the only validated biomarker for esophageal adenocarcinoma (EAC)-risk available. In an unselected BE-population the risk of developing EAC is low, 0.12% annually. In patients with BE and low-grade dysplasia (LGD) the number of EAC is 5,1 per 1000 person-years according to a large Danish cohort-study. New biomarkers are warranted for better patient selection before inclusion into BE surveillance programmes.

Epidemiologic studies have demonstrated suppressed numbers of cancer prevalence in cohorts being under different medical treatment. Anti-inflammatory, lipid-lowering and anti-hypertensive drugs are mentioned. In a British epidemiological study 2007 Sjöberg et al noted a lower prevalence of EAC among patients treated with antihypertensive drugs interfering with the renin-angiotensin system (RAS) such as AT1R-blockers and ACE-inhibitors. Wegman-Ostrosky et al linked RAS to the "Hallmarks of cancer" by RAS directly affecting tumor and stromal cells, and indirectly by affecting vascular cells in angiogenesis.

RAS is known to be involved in fluid and electrolyte homeostasis and in hemodynamic regulation. The last decade this endocrine signalling system has been proven to utilise tissue-based character, being involved in pathological conditions such as inflammation, wound-healing and even cancer, in several organ systems.

The "classical" signalling pathway of RAS, when angiotensin II (AngII) is being formed by the help of angiotensin converting enzyme (ACE) and its affinity to the membrane-bound receptors (angiotensin II type 1 and 2 receptors (AT1R and AT2R)), is now being challenged by the discovery of "alternative" pathways with enzymes and receptors, making the picture more diverse.

Reports from the investigators laboratory indicate the existence of a local RAS in the esophageal wall musculature and in the squamous mucosa. This was further explored by Björkman et al 2013, showing that some RAS-components are significantly altered in patients with erosive reflux disease when compared to healthy volunteers. In the investigators latest explorative study, the investigators discovered the altered expression of "classical" RAS components in BE with and without dysplasia (unpublished results).

By a possible alteration in RAS-related protein-expression in BE with increasing grade of dysplasia towards EAC, the investigators may have a possible "pathway" leading to biomarkers for cancer-development. Furthermore, the already well-known anti-hypertensive drugs ACE-inhibitors and AT1R-blockers may interfere with the risk of malignancy in BE. The investigators therefore wish to test, in a exploratory prospective randomized placebo-controlled setting, whether RAS-related protein-expressions in BE are altered by the addition of RAS-suppressant pharmaceuticals. In the same manner the investigator wish to see if the expressions of well-known biomarkers for cancer and inflammation are altered.

ELIGIBILITY:
Inclusion Criteria:

* Barretts esophagus with a minimum length of 1 cm and histomorphologically confirmed low grade dysplasia

Exclusion Criteria:

* Treatment with ACE-inhibitors (angiotensin converting enzyme inhibitors) or AT1R-antagonists (angiotensin type 1 receptor antagonists). Newly diagnosed or treatment resistant hypertonia or renal failure.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in expression of proteins associated with inflammation, proliferation and cancer development | Assessed at baseline (day 0) and after three weeks (day 21) of treatment
  Change in expression of p53, AMACR, Caspase 3, iNOS, VEGFR2, EGFR, CyclinD1, NFkB, PPARy, Cox-2, NLRP3 and MPO after 3 weeks treatment, assessed by Western blot.

SECONDARY OUTCOMES:
Change in regulation of potential new biomarkers associated with esophageal cancer | Assessed at baseline (day 0) and after three weeks (day 21) of treatment
  Change in regulation after 3 weeks treatment of proteins associated with esophageal cancer assessed by global proteomic analysis. Expression of regulated proteins found in the proteomic analysis are further investigated with Western blot.

CONTACTS AND LOCATIONS:
Overall Officials: Anders F Edebo, MD PhD, Study Director — Dept. of Gastrosurgical Research and Education, Inst. Clinical Sciences
Locations (1):
- Dept. of Gastrosurgical Research and Education, Inst. Clinical Sciences, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No